CLINICAL TRIAL: NCT04388514
Title: Blood Ozonization in Patients With SARS-CoV-2 Respiratory Failure
Acronym: CORMOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Collaborators: Fondazione Toscana Gabriele Monasterio (Other); Policlinico Militare, Roma - Italy (Unknown); Ospedale San Liberatore di Atri (Unknown); Ospedale Umberto I di Torino (Other); Università di Siena (Unknown); Ospedale Civile di Lucca (Unknown); Ospedale di Siracusa (Unknown); Azienda Sanitaria Locale di Vercelli (Other)
Responsible Party: Principal Investigator, Carlo Tascini, Infectious Diseases Department, Azienda Sanitaria-Universitaria Integrata di Udine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIG: Z7C2CA5837
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: SARS-CoV-2 Respiratory Failure
Keywords: SARS-CoV-2; Respiratory Failure; COVID-19; medical ozone; ozone therapy; cytokine release syndrome
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19; Cytokine Release Syndrome

STUDY DESIGN:
Intervention Model Description: The study includes 2 arms:
  * Arm A: Blood ozonization plus BAT (n= 45 subjects)
  * Arm B: Standard of Care only without Blood ozonization (n= 45 subjects)
  To note that the Standard of Care are therapy with antiretroviral therapy (lopinavir/ritonavir 2 tablets every 12 hours or darunavir/cobicistat 1 tablet per day) and hidrossycloroquine 400 mg every 12 hours then first day, followed by 200 mg every 12 hours for other 4 days
Who Masked: Investigator
Masking Description: Randomization, 1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood ozonization (Experimental): Blood ozonization plus BAT
  Interventions: Procedure: Medical Ozone procedure
- Standard of Care (No Intervention): BAT "only"
  To note that the BAT are therapy with antiretroviral therapy (lopinavir/ritonavir 2 tablets every 12 hours or darunavir/cobicistat 1 tablet per day) and hidrossycloroquine 400 mg every 12 hours then first day, followed by 200 mg every 12 hours for other 4 days.

INTERVENTIONS:
Procedure: Medical Ozone procedure — The systemic ozone treatment procedure was decided by the physician on duty and started preliminarily at the patient's bed with the drawing of autologous blood and, after proper O2/O3 mixing, with its re-infusion. After junction of an adequate venous patient's way with a dedicated latex free plastic bag containing 35 ml of sodium citrate, a blood amount of 200 ml is taken. At the end, the withdrawal line was washed and the re-infusion one was filled with saline solution. The blood, without any patient disconnection, was then mixed with a gas mixture of a 200 cc composed by 96% of Oxygen and 4% of Ozone with a therapeutic O3 range of 40 μg/mL of gas per mL of blood. In order to guarantee the O2/O3 homogeneous diffusion into the blood, the bag was gently mixed for about 10 minutes, therefore the blood was re-infused into the patients. The duration of ozone treatment lasted for 3 consecutive days.
  Arms: Blood ozonization

SUMMARY:
Aim. The emerging outbreak of coronavirus disease 2019 (COVID-19) caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) continues to spread worldwide. Beside the prescription of some promising drugs as chloroquine, azithromycin, antivirals (lopinavir/ritonavir, darunavir/cobicistat) and immunomodulating agents (steroids, tocilizumab), in our patients with mild to moderate pneumonia due to SARS-CoV-2 we planned a randomize study to evaluate, respect the best available therapy (BAT), the use of autohemotherapy treatement with an oxygen/ozone (O3) gaseous mixture as adjuvant therapy.

Design. Multicentric, randomized study.

Participants. Clinical presentations are based upon clinical phenotypes identified by the Italian Society of Emergency and Urgency Medicine (SIMEU - Società Italiana di Medicina di Emergenza-Urgenza) and patients that meet criteria of phenotypes 2 to 4 were treat with best available therapy (BAT), and randomized to receive or not O3-autohemotherapy.

Main outcome measures. The end-point were the time of respiratory improvement and earlier weaning from oxygen support: these parameters were included in the SIMEU clinical phenotypes classification.

DETAILED DESCRIPTION:
Recruitment Details.

The investigator enrolled, in the study, subjects with COVID-19 modest to moderate respiratory insufficiency (SIMEU clinical phenotypes 2-4) thus cared in an infectious disease ward.

To note that The Italian Society of Emergency and Urgency Medicine (SIMEU - Società Italiana di Medicina di Emergenza-Urgenza) suggest to classified the COVID-19 patients in 5 clinical phenotypes:

* Phenotype 1: subjects with fever and without respiratory failure (normal Arterial Blood Gas analysis - ABG -, six-minute walking test - 6mWT - and Chest XR). These patients usually can manage at home maintaining quarantine period.
* Phenotype 2: subjects with fever but with ABG and/or Chest XR indicative of modest respiratory insufficiency (PO2> 60 mmHg in ambient air) and / or pulmonary consolidation area. These patients need to be hospitalized because they can get quickly worse.
* Phenotype 3: subjects with fever associate to moderate-severe respiratory insufficiency (at triage PO2< 60 mmHg in ambient air) and /or bilateral pulmonary consolidation area at Chest XR. These patients need to be treated with high flow oxygen therapy.
* Phenotype 4: subjects with respiratory failure with suspected ARDS (Adult Respiratory Distress Syndrome) or complicated pneumonia. These patients require hospitalization in sub-intensive care unit.
* Phenotype 5: subject with ARDS at the beginning. These patients will require Intensive Care Unit (ICU) admission and non-invasive positive pressure ventilation (NIPPV) or mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Male and no pregnant female patients 18 years of age or older were eligible if they had a diagnostic specimen that was positive on RT-PCR, had pneumonia confirmed by chest imaging and gave their informed consent to participate at the study

Exclusion Criteria:

* Exclusion criteria were pregnancy, G6PHD (glucose 6 phosphate dehydrogenase) deficiency, concomitant serious disease and failure to obtain informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-10-08 (Estimated); Study Completion 2020-10-08 (Estimated)

PRIMARY OUTCOMES:
Time of respiratory improvement and earlier weaning from oxygen support | 3 days
  Evaluation of ABG paramethers the day after the last blood ozonization procedure (Day 3)
The time of respiratory improvement and earlier weaning from oxygen support | 10 days
  Evaluation of ABG paramethers the one week after the last blood ozonization procedure (Day 10)

SECONDARY OUTCOMES:
Assessment of the length of hospitalization | up to 90 days
  Asse the lenghth of hospital stay in the two arms
Assessment of the length of Intensive Care Unit (ICU) stay | up to 90 days
  Asse the lenghth of ICU stay in the two arms
Improvment in chest imaging finding | 10 days
  improving, worsening or stability of the chest imaging (chest CT, Chest XR and/or Point-of-Care Ultrasound) finding in the two arms
Improvment in cytokine release syndrome | 10 days
  Evaluation of plasmatic cytochine (IL-6, lymphocyte typing for CD4, CD3, CD8, HLA-DR, CD45) response in the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Amato De Monte, Study Chair — Presidio Ospedaliero Universitario "Santa Maria della Misericordia", Udine - Italy
Locations (1):
- Dott. Amato De Monte, Udine, Italy

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: Contacting the Principal Investigator

REFERENCES:
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Elvis AM, Ekta JS. Ozone therapy: A clinical review. J Nat Sci Biol Med. 2011 Jan;2(1):66-70. doi: 10.4103/0976-9668.82319. PMID 22470237
- [Background] Bocci VA. Scientific and medical aspects of ozone therapy. State of the art. Arch Med Res. 2006 May;37(4):425-35. doi: 10.1016/j.arcmed.2005.08.006. PMID 16624639
- [Background] Smith NL, Wilson AL, Gandhi J, Vatsia S, Khan SA. Ozone therapy: an overview of pharmacodynamics, current research, and clinical utility. Med Gas Res. 2017 Oct 17;7(3):212-219. doi: 10.4103/2045-9912.215752. eCollection 2017 Jul-Sep. PMID 29152215
- [Background] Gulmen S, Kurtoglu T, Meteoglu I, Kaya S, Okutan H. Ozone therapy as an adjunct to vancomycin enhances bacterial elimination in methicillin resistant Staphylococcus aureus mediastinitis. J Surg Res. 2013 Nov;185(1):64-9. doi: 10.1016/j.jss.2013.05.085. Epub 2013 Jun 19. PMID 23809152
- See also: SIMEU Classification and Guidelines — https://www.simeu.it/w/articoli/leggiArticolo/3964/leggi
- See also: doi: 10.4081/ozone.2020.9014. — https://www.pagepressjournals.org/index.php/ozone/article/view/9014

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT04388514/Prot_SAP_000.pdf